CLINICAL TRIAL: NCT02784275
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Evaluate the Efficacy and Safety of Cyclo-Z in Patients With Obese Type 2 Diabetes
Brief Title: A Study to Evaluate the Efficacy and Safety of Cyclo-Z in Patients With Obese Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovMetaPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMP-CYZ-P2-001
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus Type 2 in Obese
MeSH Terms: interventions — Z 008

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose A (Experimental): Cyclo-Z containing 23 mg zinc plus 3 mg CHP
  Interventions: Drug: Cyclo-Z
- Dose B (Experimental): Cyclo-Z containing 23 mg zinc plus 9 mg CHP
  Interventions: Drug: Cyclo-Z
- Dose C (Experimental): Cyclo-Z containing 23 mg zinc plus 15 mg CHP
  Interventions: Drug: Cyclo-Z
- Dose D (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclo-Z
  Arms: Dose A; Dose B; Dose C
Drug: Placebo
  Arms: Dose D

SUMMARY:
This is a double-blind, randomized, placebo-controlled, parallel-group comparison study to evaluate the efficacy and safety of Cyclo-Z for the treatment of subjects with obese type 2 diabetes.

The study will consist of 3 phases:

* Screening phase (2 weeks)
* Treatment phase (12 weeks)
* Follow-up phase (2 weeks)

Following a 2-week screening period, subjects who meet all inclusion and exclusion criteria will be randomly assigned into one of the following treatment arms:

* Dose A: Cyclo-Z containing 23 mg zinc plus 3 mg CHP - 16 subjects
* Dose B: Cyclo-Z containing 23 mg zinc plus 9 mg CHP - 16 subjects
* Dose C: Cyclo-Z containing 23 mg zinc plus 15 mg CHP - 16 subjects
* Dose D: Placebo - 16 subjects

The assigned dose will be orally administered to subjects once a day before bedtime for 12 consecutive weeks. After the randomization at Week 0 (Visit 2), subjects will visit their respective trial sites at Weeks 2, 4, 6, 8, 10, 12, and 14 (Visits 3, 4, 5, 6, 7, 8, and 9).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 or older.
2. Subjects diagnosed with type 2 diabetes mellitus according to the American Diabetes Association (ADA) criteria.
3. Subjects treated with stable doses of insulin and/or other hypoglycemic agent(s) for type 2 diabetes mellitus for at least 2 months prior to randomization.
4. Subjects whose fasting blood glucose levels are reasonably stable for at least 2 months prior to randomization and during the 2-week screening period.
5. Subjects who have Hemoglobin A1c levels of 7.5 to 10.0 % at Screening.
6. Subjects whose BMI is 30 or above.
7. Subjects who can give written informed consent.

Exclusion Criteria:

1. Subjects who have any DM-related end-organ damages.
2. Subjects who have a history of diabetic ketoacidosis or hyperosmolar non-ketotic coma.
3. Subjects who have any disease likely to limit life span and/or increase risks of interventions such as:

   * Carotid B-mode ultrasound test results indicating clinically significant stenosis in the common carotid arteries requiring intervention by angioplasty or resection.
   * Cancer treatment in the past 5 years, with the exception of cancers which have been cured, and carry a good prognosis.
   * Infectious disease: HIV positivity, active tuberculosis, or pneumonia.
4. Subjects who have any of the following conditions related to cardiovascular disease:

   * Hospitalization for the treatment of heart disease in the past 12 months.
   * New York Heart Association Functional Class > 2.
   * Left Bundle branch block on ECG at Screening.
   * Third degree atrioventricular block on ECG at Screening.
   * Uncontrolled hypertension with average systolic blood pressure of > 160 mmHg or diastolic blood pressure > 95 mmHg at Screening and Baseline.
   * Pulse rate > 95 beats per minute at Screening and Baseline.
   * Stroke or transient ischemic attack in the past 12 months.
5. Subjects who have any of the following conditions related to gastrointestinal disease:

   * Chronic hepatitis or cirrhosis.
   * Episode of alcoholic hepatitis or alcoholic pancreatitis in the past 2 months.
   * Inflammatory bowel disease requiring treatment in the past 12 months.
   * Significant abdominal surgery (e.g., gastrectomy, gastric bypass) in the past 2 months.
6. Subjects who have serum creatinine > 1.5 mg/dL for male or > 1.4 mg/dL for female.
7. Subjects who have chronic obstructive airway disease or asthma requiring daily therapy or home use oxygen.
8. Subjects who have hematocrit < 36.0% for male or < 33.0% for female.
9. Subjects who have any of the following conditions or behaviors likely to affect the conduct of the study:

   * Weight loss of > 10% in the past 6 months.
   * Unable to walk without assisted device.
   * Major psychiatric disorder which would impede conduct of the research.
   * Excessive alcohol intake (i.e., more than 2 drinks/day).
10. Subjects who take any of the following medications:

    * Psychoactive agents such as monoamine oxidase inhibitors and antidepressants (e.g., lithium, Prozac, Zoloft, Serzone, Paxil, Effexor).
    * Any other medications that may pose harm to the subject.
11. Female subjects who have a positive serum pregnancy test at Screening, plan a pregnancy during study period, or are breast feeding.
12. Female subjects who don't meet any of the following criteria:

    * Surgically sterile (i.e., have had bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) at least 6 months before randomization.
    * Post-menopausal for at least 12 months prior to Screening.
    * If sexually active, they should use oral contraceptives, double barrier contraception (e.g., condom with spermicide), intrauterine device, or other methods approved by the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Lee, Study Director — KCRN Research
Locations (4):
- United States (4):
  - Los Angeles, California
  - Hialeah, Florida
  - Houston, Texas
  - Tomball, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 mg CHP Plus 23 mg Zinc: Cyclo-Z containing 23 mg zinc plus 3 mg CHP
  Cyclo-Z
- 9 mg CHP Plus 23 mg Zinc: Cyclo-Z containing 23 mg zinc plus 9 mg CHP
  Cyclo-Z
- 15 mg CHP Plus 23 mg Zinc: Cyclo-Z containing 23 mg zinc plus 15 mg CHP
  Cyclo-Z
- Placebo: Placebo
  Placebo
Period: Overall Study
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Started | 16 | 16 | 17 | 15
Completed | 15 | 16 | 16 | 14
Not Completed | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 17 | 15 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 15 | 14 | 54
  >=65 years | 2 | 5 | 2 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of the subjects at the time of study entry.
  years | 56.9 (7.58) | 59.9 (9.89) | 55.2 (10.90) | 57.1 (5.53) | 57.3 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 8 | 28
  Male | 11 | 9 | 9 | 7 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 4 | 5 | 24
  Not Hispanic or Latino | 10 | 7 | 13 | 9 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 17 | 15 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change of HbA1c Level From Baseline
Description: Change in HbA1c from Day 1 to Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However only 54 subjects had Week 12 values (12, 15, 14, and 13 subjects, respectively).
Measure: Mean (Standard Deviation); unit: (%)
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 15 | 14 | 13
(%) | -0.21 (0.979) | -0.17 (1.038) | -0.43 (1.132) | -0.04 (1.068)

2. Primary Outcome: Change of Body Weight From Baseline
Description: Change in body weight from Day 1 to Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 54 subjects had Week 12 values for weight (12, 15, 14, and 13, respectively).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 15 | 14 | 13
kg | -0.73 (1.524) | 0.61 (3.4) | -0.92 (2.381) | 2.38 (5.702)

3. Secondary Outcome: Change of Fasting Plasma Glucose Level From Baseline
Description: Change in fasting plasma glucose from Day 1 to Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 54 subjects had Week 12 values (12, 15, 14, and 13, respectively).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 15 | 14 | 13
mg/dL | -10.4 (59.20) | 25.4 (65.66) | 5.3 (49.24) | -23.4 (95.78)

4. Secondary Outcome: Proportion of Subjects Achieving HbA1c Goal of <7.0%
Description: Percent of subjects who achieved HbA1c of <7% at Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 54 subjects had Week 12 values (12, 15, 14, and 13 respectively).
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 15 | 14 | 13
Participants | 4 | 3 | 2 | 2

5. Secondary Outcome: Proportion of Subjects Achieving HbA1c Goal of <6.5%
Description: Percent of subjects who achieved HbA1c of <6% at Week 12
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 15 | 14 | 13
Participants | 0 | 0 | 1 | 1

6. Secondary Outcome: Change in Waist Circumference From Baseline
Description: Change in waist circumference from Day 1 to Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 53 subjects had Week 12 values (12, 14, 14, and 13 respectively).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 14 | 14 | 13
cm | -0.71 (6.881) | -1.31 (4.099) | -0.70 (8.812) | -0.79 (5.144)

7. Secondary Outcome: Change of Postprandial (2 Hours After Dinner) Blood Glucose Level From Baseline
Description: Change in postprandial (2 hours after dinner) blood glucose levels from Day 1 to Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 51 subjects had Week 12 postprandial glucose values (11, 14, 14, and 12, respectively).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 11 | 14 | 14 | 12
mg/dL | -14.56 (40.210) | 8.78 (38.543) | -5.25 (62.754) | -13.95 (54.262)

8. Secondary Outcome: Change of Oral Glucose Tolerance Test From Baseline
Description: Change in oral glucose tolerance test results from Day 1 to Week 12
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 53 subjects had Week 12 oral glucose tolerance test results (12, 15, 14, and 12, respectively).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 12 | 15 | 14 | 12
mg/dL | -13.8 (51.16) | 28.4 (89.45) | -19.6 (85.62) | -33.6 (75.72)

9. Secondary Outcome: Change of Score in Audit of Diabetes-Dependent Quality of Life Questionnaire From Baseline
Description: Individual 19 domains were calculated as a weighted score (WS) for each domain. Average weighted impact score = summing of WS for each domain/19 domains. Total range possible is -9 to 3, and higher number means improvement in quality of life.
Time Frame: 12 weeks
Population: Efficacy Analysis Set (N=61) was used for the efficacy analysis. However, only 51 subjects had Week 12 ADDQoL results (9, 15, 14, and 13, respectively).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
Number analyzed (Participants) | 9 | 15 | 14 | 13
Score on a scale | -0.23 (2.311) | 0.21 (2.171) | 0.35 (1.075) | 1.53 (2.655)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | 3 mg CHP Plus 23 mg Zinc | 9 mg CHP Plus 23 mg Zinc | 15 mg CHP Plus 23 mg Zinc | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/16 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 5/15 | 7/16 | 13/16 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg CHP Plus 23 mg Zinc (N=15) | 9 mg CHP Plus 23 mg Zinc (N=16) | 15 mg CHP Plus 23 mg Zinc (N=16) | Placebo (N=14)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg CHP Plus 23 mg Zinc (N=15) | 9 mg CHP Plus 23 mg Zinc (N=16) | 15 mg CHP Plus 23 mg Zinc (N=16) | Placebo (N=14)
Blood glucose increased (Investigations) | 1 (1) | 4 (5) | 4 (5) | 1 (2)
Blood insulin increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Blood zinc increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Glucose urine present (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haemotocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT02784275/SAP_000.pdf
  • Study Protocol (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT02784275/Prot_001.pdf